CLINICAL TRIAL: NCT03902418
Title: Evaluation of Pre-Exposure Prophylaxis (PrEP) Initiation, Retention, and Adherence in Pregnant and Breastfeeding Women
Brief Title: Evaluation of Pre-Exposure Prophylaxis (PrEP) in Pregnant and Breastfeeding Women
Acronym: PrEP-PP
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Principal Investigator, University of California, Los Angeles
Other Study IDs: 1R01MH116771-01A1 (NIH)
Record Dates: First submitted 2019-01-10; First posted 2019-04-04 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: HIV-I Infection
Keywords: Prevention in Pregnant and Breastfeeding Women; HIV Pre-Exposure Prophylaxis (PrEP)
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: emtricitabine/tenofovir — Women recruited at ante-natal clinics, counseled about PrEP, and provided medication and follow up if desired
  Other Names: Behavioral Counseling

SUMMARY:
The investigators will conduct an observational cohort study in 1200 pregnant women who will be recruited at the first antenatal care (ANC) visit from the Gugulethu and one additional facility in the Klipfontein-Mitchell's Plain subdistrict of the Metro Region (to be identified in conjunction with provincial and local health authorities) Midwife Obstetric Units in Cape Town (n=600 pregnant women per site). The enrolled women will be followed through 12-months post-delivery.

DETAILED DESCRIPTION:
The objectives of the study are to:

1. Determine the distribution of women across the PrEP cascade:

1. Evaluate the proportion of pregnant and breastfeeding women who initiate PrEP out of all women offered PrEP
2. Evaluate the proportion of pregnant and breastfeeding women who are retained in the PrEP cohort
3. Evaluate the proportion of pregnant and breastfeeding women who initiate PrEP who adhere to PrEP using objective dried blood spot measures and subjective measures of self-reported pill count and adherence
4. Evaluate the proportion of pregnant and breastfeeding women on PrEP (and not on PrEP) who acquire HIV, who transmit HIV to their infant, and who report adverse events 2. Evaluate patient and provider-level factors associated with the PrEP cascade using quantitative and qualitative approaches (including in-depth interviews) 3. Apply an established mathematical model to simulate the impact of improvement in the PrEP cascade on HIV infections averted (maternal and perinatal)

ELIGIBILITY:
Inclusion Criteria:

* >16 years of age,
* confirmed HIV-negative (using 2 rapid tests,
* confirmed with a 4th generation antigen HIV test;
* lives within 20 km. of the clinic;
* confirmed to be pregnant;
* without psychiatric or medical contraindications to PrEP

Exclusion Criteria:

* Concurrent enrollment in another HIV-1 vaccine or prevention trial;
* medical hospitalization in the past year for any reason;
* receipt of TB treatment in the past 30 days; history of renal disease;
* exhibiting psychotic symptoms (including hallucinations, suicidal or homicidal ideation, or violent behavior),
* currently or history of taking anti-psychotic medications;
* positive Hepatitis B surface antigen test on screening;
* history of bone fracture not related to trauma;
* any other medical, psychiatric, or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study.

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Study counselors will enroll consecutive eligible, consenting pregnant adolescent girls (>16 years) and women in ANC (n=600 women per site; N=1200 pregnant women) and follow them up for 12-months postpartum or until censorship for a mean of 18-months' follow-up.
  In a sub-study, STI and PrEP in Pregnancy Study (STIPPS), we will include n=268 women who recieve point of care STI results vs. those treated syndromically to evaluate PrEP initiation in pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MD PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Background] Joseph Davey DL, Daniels J, Beard C, Mashele N, Bekker LG, Dovel K, Ncayiyana J, Coates TJ, Myer L. Healthcare provider knowledge and attitudes about pre-exposure prophylaxis (PrEP) in pregnancy in Cape Town, South Africa. AIDS Care. 2020 Oct;32(10):1290-1294. doi: 10.1080/09540121.2020.1782328. Epub 2020 Jun 23. PMID 32576023
- [Result] Joseph Davey DL, Wilkinson L, Grimsrud A, Nelson A, Gray A, Raphael Y, Wattrus C, Pillay Y, Bekker LG. Urgent appeal to allow all professional nurses and midwives to prescribe pre-exposure prophylaxis (PrEP) in South Africa. S Afr Med J. 2023 Aug 3;113(8):12-16. doi: 10.7196/SAMJ.2023.v113i8.1191. No abstract available. PMID 37882113
- [Result] Khadka N, Gorbach PM, Nyemba DC, Mvududu R, Mashele N, Javanbakht M, Nianogo RA, Aldrovandi GM, Bekker LG, Coates TJ, Myer L, Joseph Davey DL. Evaluating the use of oral pre-exposure prophylaxis among pregnant and postpartum adolescent girls and young women in Cape Town, South Africa. Front Reprod Health. 2023 Sep 19;5:1224474. doi: 10.3389/frph.2023.1224474. eCollection 2023. PMID 37795521
- [Result] Li KT, Li F, Jaspan H, Nyemba D, Myer L, Aldrovandi G, Joseph-Davey D. Changes in the Vaginal Microbiome During Pregnancy and the Postpartum Period in South African Women: a Longitudinal Study. Reprod Sci. 2024 Jan;31(1):275-287. doi: 10.1007/s43032-023-01351-4. Epub 2023 Sep 18. PMID 37721699
- [Result] Haribhai S, Khadka N, Mvududu R, Mashele N, Bekker LG, Gorbach P, Coates TJ, Myer L, Joseph Davey DL. Psychosocial determinants of pre-exposure prophylaxis use among pregnant adolescent girls and young women in Cape Town, South Africa: A qualitative study. Int J STD AIDS. 2023 Jul;34(8):548-556. doi: 10.1177/09564624231152776. Epub 2023 Mar 22. PMID 36947792
- [Result] Joseph Davey D, Nyemba DC, Castillo-Mancilla J, Wiesner L, Norman J, Mvududu R, Mashele N, Johnson LF, Bekker LG, Gorbach P, Coates TJ, Myer L. Adherence challenges with daily oral pre-exposure prophylaxis during pregnancy and the postpartum period in South African women: a cohort study. J Int AIDS Soc. 2022 Dec;25(12):e26044. doi: 10.1002/jia2.26044. PMID 36480171
- [Result] Joseph Davey D, Hsiao NY, Wendy Spearman C, Sonderup M, Hu NC, Mashele N, Mvududu R, Myer L. Low prevalence of hepatitis B virus infection in HIV-uninfected pregnant women in Cape Town, South Africa: implications for oral pre-exposure prophylaxis roll out. BMC Infect Dis. 2022 Sep 1;22(1):719. doi: 10.1186/s12879-022-07697-5. PMID 36050648
- [Result] Beesham I, Mansoor LE, Joseph Davey DL, Palanee-Phillips T, Smit J, Ahmed K, Selepe P, Louw C, Singata-Madliki M, Kotze P, Heffron R, Parikh UM, Wiesner L, Rees H, Baeten JM, Beksinska M. Brief Report: Quantifiable Plasma Tenofovir Among South African Women Using Daily Oral Pre-exposure Prophylaxis During the ECHO Trial. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):26-30. doi: 10.1097/QAI.0000000000003023. Epub 2022 Jun 9. PMID 35972853
- [Result] Miller AP, Shoptaw S, Mvududu R, Mashele N, Coates TJ, Bekker LG, Essack Z, Groenewald C, Petersen Z, Gorbach PM, Myer L, Joseph Davey DL. Sexual Risk among Pregnant Women at Risk of HIV Infection in Cape Town, South Africa: What Does Alcohol Have to Do with It? AIDS Behav. 2023 Jan;27(1):37-50. doi: 10.1007/s10461-022-03742-1. Epub 2022 Jun 23. PMID 35737280
- [Result] Beesham I, Dovel K, Mashele N, Bekker LG, Gorbach P, Coates TJ, Myer L, Joseph Davey DL. Barriers to Oral HIV Pre-exposure Prophylaxis (PrEP) Adherence Among Pregnant and Post-partum Women from Cape Town, South Africa. AIDS Behav. 2022 Sep;26(9):3079-3087. doi: 10.1007/s10461-022-03652-2. Epub 2022 Mar 22. PMID 35316471
- [Result] Joseph Davey DL, Mvududu R, Mashele N, Lesosky M, Khadka N, Bekker LG, Gorbach P, Coates TJ, Myer L. Early pre-exposure prophylaxis (PrEP) initiation and continuation among pregnant and postpartum women in antenatal care in Cape Town, South Africa. J Int AIDS Soc. 2022 Feb;25(2):e25866. doi: 10.1002/jia2.25866. PMID 35138678
- [Result] Joseph Davey DL, Dovel K, Mvududu R, Nyemba D, Mashele N, Bekker LG, Gorbach PM, Coates TJ, Myer L. Pre-exposure Prophylaxis Recent Adherence With Real-Time Adherence Feedback and Partner Human Immunodeficiency Virus Self-Testing: A Pilot Trial Among Postpartum Women. Open Forum Infect Dis. 2021 Dec 23;9(2):ofab609. doi: 10.1093/ofid/ofab609. eCollection 2022 Feb. PMID 35097151
- [Result] Joseph Davey DL, Bekker LG, Bukusi EA, Chi BH, Delany-Moretlwe S, Goga A, Lyerly AD, Mgodi NM, Mugo N, Myer L, Noguchi LM, Stranix-Chibanda L, Slack C, Pintye J. Where are the pregnant and breastfeeding women in new pre-exposure prophylaxis trials? The imperative to overcome the evidence gap. Lancet HIV. 2022 Mar;9(3):e214-e222. doi: 10.1016/S2352-3018(21)00280-0. Epub 2022 Jan 25. PMID 35090604
- [Result] Moran A, Mashele N, Mvududu R, Gorbach P, Bekker LG, Coates TJ, Myer L, Joseph Davey D. Maternal PrEP Use in HIV-Uninfected Pregnant Women in South Africa: Role of Stigma in PrEP Initiation, Retention and Adherence. AIDS Behav. 2022 Jan;26(1):205-217. doi: 10.1007/s10461-021-03374-x. Epub 2021 Jul 21. PMID 34287756
- [Result] Joseph Davey DL, Knight L, Markt-Maloney J, Tsawe N, Gomba Y, Mashele N, Dovel K, Gorbach P, Bekker LG, Coates TJ, Myer L. "I had Made the Decision, and No One was Going to Stop Me" -Facilitators of PrEP Adherence During Pregnancy and Postpartum in Cape Town, South Africa. AIDS Behav. 2021 Dec;25(12):3978-3986. doi: 10.1007/s10461-021-03320-x. Epub 2021 Jun 3. PMID 34085132
- [Derived] de Voux A, Nyemba DC, Silliman M, Mashele N, Mvududu R, Myer L, Joseph Davey D. Point-of-care testing for sexually transmitted infections and HIV pre-exposure prophylaxis among pregnant women in South Africa, 2021-2022: randomised controlled trial. Sex Transm Infect. 2024 Feb 19;100(2):77-83. doi: 10.1136/sextrans-2023-055975. PMID 38124133

RESULTS

PARTICIPANT FLOW:
Groups:
- PrEP Use: Evaluation of PrEP use among pregnant and breastfeeding women including initiation, continuation and adherence (self report and objective outcomes)
Period: Overall Study
Arm/Group | PrEP Use
Started | 1195
Completed | 1092
Not Completed | 103

BASELINE CHARACTERISTICS:
Population: Pregnant women in PrEP-PP study
Arm/Group | PrEP Use
Number analyzed (Participants) | 1195
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1195
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1195
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 1195

OUTCOME MEASURES:

1. Primary Outcome: Participants Initiating Pre-exposure Prophylaxis During Pregnancy
Description: Percentage of participants initiating pre-exposure prophylaxis during pregnancy
Time Frame: Percentage of participants initiating pre-exposure prophylaxis between first ante-natal clinic visit and birth of infant
Measure: Count of Participants; unit: Participants
Groups:
- Pregnant Women Initiating PrEP: Pregnant women in antenatal care (16+ years) who initiated PrEP among all women who were offered oral TDF/FTC as PrEP in a cohort study
Arm/Group | Pregnant Women Initiating PrEP
Number analyzed (Participants) | 1195
Participants | 1089

2. Primary Outcome: Adherence to TDF at 3-months on PrEP
Description: Percentage of participants with red blood cells with >80% levels at >40ng/mL TDF-DP at 3 months on PrEP
Time Frame: Measured at 3 month follow up visit
Population: 382 women on PrEP with dried blood spots measured for TFV-DP
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Initiating PrEP
Number analyzed (Participants) | 382
Participants | 256

3. Primary Outcome: Women Initiating Pre-exposure Prophylaxis Post-partum
Description: Percentage of women initiating pre-exposure prophylaxis
Time Frame: Percentage of participants initiating pre-exposure prophylaxis at first post-partum to final post-partum visit 12 months after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Initiating PrEP
Number analyzed (Participants) | 1195
Participants | 1009

4. Primary Outcome: Adherence to TDF at 6 Months Post-partum
Description: Percentage of participants with red blood cells with >80% levels at >40ng/mL TDF-DP at 6 month post-partum visit
Time Frame: Measured at 6-month post-partum visit
Population: Women with TFV-DP in DBS at 6m visit
Measure: Count of Participants; unit: Participants
Groups:
- Women With Quantifiable Adherence to TFV-DP at 6-month Visit: Pregnant women in antenatal care (16+ years) with quantifiable TFV-DP levels (any vs none) among those offered oral TDF/FTC as PrEP and reporting taking PrEP in the last 30-days at 6-months
Arm/Group | Women With Quantifiable Adherence to TFV-DP at 6-month Visit
Number analyzed (Participants) | 175
Participants | 51

5. Primary Outcome: Number of Participants With Adherence to TFV-DP at 6-month Visit
Description: Quantifiable TFV (versus none) using dried blood spots (DBS) taken at 6-month study visit among subset of women who reported taking PrEP in the last 30-days at 6-months
Time Frame: Measured at 6-month study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Women With Quantifiable Adherence to TFV-DP at 6-month Visit
Number analyzed (Participants) | 186
Participants | 86

6. Secondary Outcome: PrEP Initiation Among Those With STI POC Testing vs Syndromic Management
Description: Proportion of those with POC (point of care) STI vs syndromic management who initiate oral PrEP
Time Frame: Measured at enrollment and 1 month follow up
Measure: Count of Participants; unit: Participants
Groups:
- Women Receiving POC STI Testing: Pregnant or postpartum women randomized to receive POC STI testing
- Women Receiving STI Syndromic Management: Pregnant or postpartum women randomized to receive STI syndromic management
Arm/Group | Women Receiving POC STI Testing | Women Receiving STI Syndromic Management
Number analyzed (Participants) | 133 | 135
Participants | 89 | 84

ADVERSE EVENTS:
Time Frame: Between Aug 2019 and October 2021, we followed 1195 women and ascertained 1145 pregnancy outcomes, abstracted from maternal case files, infant road to health cards, and local obstetric records.
Description: Miscarriage or pregnancy loss was defined as noninduced pregnancy loss ≤20 weeks (0/7 days) of gestation.
  Stillbirth was defined as delivery of a baby with no sign of life >20 weeks (0/7 days) of gestation, including foetal demise.
  Neonatal mortality was defined as death of a newborn in the first 28 days of life (days 0-27).
  Preterm live birth was defined as birth before completion of 37 weeks (0/7 days) of gestation.
  Low birthweight was defined as an infant birthweight <2500 grams.
Groups:
- Pregnant Women Offered PrEP: Pregnant women in antenatal care (16+ years) were offered oral TDF/FTC as PrEP in a cohort study
Arm/Group | Pregnant Women Offered PrEP
All-Cause Mortality (participants affected / at risk) | 0/1195
Serious Adverse Events (participants affected / at risk) | 67/1195
Other Adverse Events (participants affected / at risk) | 201/1082
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pregnant Women Offered PrEP (N=1195)
Pregnancy Loss, Miscarriage (Pregnancy, puerperium and perinatal conditions) | 36/1145 — Miscarriages occurring at gestational age <= 20 weeks among participants with available pregnancy outcomes
Pregnancy Loss, Stillbirth (Pregnancy, puerperium and perinatal conditions) | 25/1145 — Stillbirth occurring at gestational age > 20 weeks among women with available pregnancy outcomes
Live Birth Outcome, Neonatal Death (Pregnancy, puerperium and perinatal conditions) | 6/1082 — Neonatal deaths observed among women with available pregnancy outcomes
HIV sero-conversion (Infections and infestations) | 16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregnant Women Offered PrEP (N=1082)
Live Birth Outcome, Preterm Delivery (Pregnancy, puerperium and perinatal conditions) | 91 — Pre-term delivery (gestational age < 37 weeks) among women with available pregnancy outcome
Live Birth Outcome, Low Birth Weight (Pregnancy, puerperium and perinatal conditions) | 110 — Low infant birth weight (<2500g) recorded among women with available pregnancy outcome

LIMITATIONS AND CAVEATS:
We originally indicated reporting "Participants Missing Pre-natal Visit" as a Secondary Outcome, however are unable to report as the data is unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03902418/Prot_SAP_ICF_000.pdf